CLINICAL TRIAL: NCT05649267
Title: Using Energy Availability as a Strategy to Explore the Effects of Relative Energy Deficiency in Sport (RED-S) on Athletes' Physiological Function, Health, and Performance
Brief Title: Using Energy Availability as a Strategy to Explore the Effects of Relative Energy Deficiency in Sport on Athletes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chen Ming You (Other)
Responsible Party: Sponsor-Investigator, Chen Ming You, student, National Taiwan Sport University
Organization: National Taiwan Sport University (Other)
Other Study IDs: IRB-3-R-026-1.1
Record Dates: First submitted 2022-11-23; First posted 2022-12-14 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Relative Energy Deficiency in Sport
MeSH Terms: conditions — Relative Energy Deficiency in Sport

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this type of study:clinical trial is to test, compare etc. In describe participant population health conditions. Participants will diet record,maintain training and life.

DETAILED DESCRIPTION:
Relative energy deficiency in sport (RED-S) can negatively affect the health and performance of both male and female athletes. The underlying etiology of RED-S is low energy availability (LEA), which occurs when there is insufficient dietary energy intake to meet exercise energy expenditure. This syndrome refers to impaired physiological function, including metabolic rate, menstrual function, bone health, immunity, protein synthesis, and cardiovascular health. Strategies to support athlete health and training energy availability are an integral part of optimizing training outcomes and preparing for competition. This project aims to investigate the prevalence of RED-S among Taiwanese athletes by recruiting athletes of different age groups and to find the relevance of dietary risk factors to enhance energy availability. This project intends to recruit athletes in aesthetic sports and weight-sensitive sports to study the prevalence of RED-S in different training periods, and to find out the relationship between the possible dietary risk factors and the improvement of energy availability, and to understand whether the strategy of improving energy availability through the concept of nutritional supplements has a positive effect on the relative energy deficiency of athletes. In the first year of this study, the prevalence of relative energy deficits, dietary risk factors in pre-season, competition and off-season will be studied for aesthetic sport and weight-sensitive sport athletes, and relevant biological indicators will be searched. In the second year of this study, the effect of carbohydrates and proteins or specific nutrients as energy availability strategies on low energy availability animal physiological function, exercise performance and overall health status will be investigated. In the third year of this sudy, the effects of carbohydrate and protein supplementation with specific nutrients as energy availability strategies on athletes' physical function, athletic performance, and overall health status during high-relative energy-deficient training will be explored. It is hoped that through the successful implementation of this research project, the results can be applied to personalized dietary planning and ensure that minimizing adverse risk factors for athletes during critical periods, which is the most important key to maintaining good health, performing at their best in training and competition, and winning the highest honor for their country on the playing field.

Keywords: Energy availability, Relative energy deficiency in sport, Low energy availability risk factors, Carbohydrate availability, Protein availability

ELIGIBILITY:
Inclusion Criteria:

* In the past year, the daily training frequency is ≥4 times/week, and each time is at least 2 hours, and there are specific special trainers

Exclusion Criteria:

* smoke

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Judoka
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2022-05-09 (Actual); Primary Completion 2023-05-09 (Estimated); Study Completion 2023-08-09 (Estimated)

PRIMARY OUTCOMES:
Body Composition Analysis | 2022/10/29~2023/07/29
  DEXA:bone mass density
DEXA:Fat Free Mass | 2022/10/29~2023/07/29
  Body Bone Composition Analysis
Inbody:Fat Free Mass | 2022/10/29~2023/07/29
  Body Composition Analysis
Inbody:Skeletal Muscle Mass. | 2022/10/29~2023/07/29
  Body Composition Analysis
Inbody:Body Fat Mass | 2022/10/29~2023/07/29
  Body Composition Analysis
Inbody:body weight | 2022/10/29~2023/07/29
  Body Composition Analysis
4 days diet record | 2022/10/29~2023/07/29
  Diet Record
Diet Recordcaculate Energy Intake. | 2022/10/29~2023/07/29
  Diet Record

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan Sport University, Taoyuan District, Taiwan